CLINICAL TRIAL: NCT00763308
Title: Fast Track Program to Create a Web-Based Cardiovascular Intervention for the Workplace
Brief Title: A Web-Based Cardiovascular Intervention for the Workplace
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Diane K. Deitz, PhD, ISA Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 535; R44HL087540-01 (NIH)
Record Dates: First submitted 2008-09-25; First posted 2008-09-30 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Cardiovascular Diseases
Keywords: Weight; Blood Pressure; Smoking Status; Cardiovascular Risk Profile
MeSH Terms: conditions — Cardiovascular Diseases; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will use the Web-based Heart Healthy program.
  Interventions: Behavioral: Web-based Heart Healthy Program
- 2 (No Intervention): Participants will receive treatment as usual.

INTERVENTIONS:
Behavioral: Web-based Heart Healthy Program — The Heart Healthy program will be developed during the course of the study based on goals set by researchers and based on feedback from focus groups. The goals of the program are to educate users in the fundamentals of heart health and risk factors for heart disease and to provide a system for starting and sustaining lifestyle changes that reduce risk of heart disease.
  Arms: 1

SUMMARY:
Heart disease is the leading cause of death in the United States, accounting for approximately 700,000 deaths a year. Heart disease can take many forms, including heart attacks, coronary artery disease, aneurysms, high blood pressure, and strokes. However, people can change things in their life to reduce the risk of getting heart disease. This study will first create an Internet-based program to help teach people about reducing heart disease risk and will then test the program in a workplace setting.

DETAILED DESCRIPTION:
Heart disease, or cardiovascular disease, refers to a range of diseases including coronary artery disease, heart attack, heart failure, high blood pressure, and stroke. These diseases are all related to problems with the heart and blood vessels, and collectively are the leading cause of death in the United States. Heart attacks or coronary artery disease sometimes have warning signs, but both can occur without warning. Approximately half of all heart attacks are fatal. Forty percent of all deaths in the United States are the result of heart disease.

Certain factors can predict whether people get heart disease. Some of these factors, like biological sex or genes inherited from a person's family, cannot be changed, but many others can. Not smoking, eating well, exercising regularly, and maintaining a healthy weight are some of the things people can do to lower their risk of heart disease. This study will develop and then test an Internet-based program that teaches people about heart health and supports them in changing behaviors that put them at risk for heart disease.

This study will be divided into two phases. In the first phase, researchers will create the Heart Healthy program, show it to focus groups, and try to improve it based on their comments. The goals of the program are to educate users in the fundamentals of heart health and risk factors for heart disease and to provide a system for starting and sustaining lifestyle changes that reduce risk of heart disease. The program will be designed for employee use in a workplace, and a tool kit will be developed for managers to supplement the employee program. The prototype will include modified segments from existing Web-based programs created by a non-profit organization, the ISA Group. The design of the program will be guided by feedback from employees and managers who use it and from experts in cardiology and epidemiology.

In the second phase, the program will be tested in a work site. Employees at risk for heart disease will be recruited and randomly assigned to receive either the Healthy Heart program or treatment as usual. Before and after the intervention, participants will be assessed on knowledge gained, attitudes changed, alterations in health behavior, and reductions in cardiovascular risk. Managers who receive the supplementary program will be tested in knowledge gained and plans for policy or procedural changes. The ultimate goal of this phase is to fully develop the Healthy Heart program for use in industry and health care settings.

ELIGIBILITY:
Inclusion Criteria:

* Works in participating company
* At least one cardiovascular risk factor

Exclusion Criteria:

* No known cardiovascular risks

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Change in health attitudes and behaviors | Measured pre- and post-intervention

SECONDARY OUTCOMES:
Change in cardiovascular risk status | Measured pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Diane K. Deitz, PhD, Principal Investigator — ISA Associates
Locations (1):
- ISA Associates, Inc., Alexandria, Virginia, United States